CLINICAL TRIAL: NCT03583476
Title: The Impact of Antibiotics MIC Value on the Efficacy of Treatment Regimens for Helicobacter Pylori Infection.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201804076RIND
Record Dates: First submitted 2018-06-22; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Resistance; Minimal inhibitory concentration; Treatment efficacy
MeSH Terms: interventions — Proton Pump Inhibitors; Metronidazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CLA triple therapy: Patients with clarithromycin-containing triple therapy
  Interventions: Drug: Proton pump inhibitor,clarithromycin,amoxicillin or metronidazole
- MET triple therapy: Patients with metronidazole-containing triple therapy
  Interventions: Drug: Proton pump inhibitor,clarithromycin,amoxicillin or metronidazole
- Concomitant therapy: Patients with concomitant therapy
  Interventions: Drug: Proton pump inhibitor,clarithromycin,amoxicillin or metronidazole
- Sequential therapy: Patients with sequential therapy
  Interventions: Drug: Proton pump inhibitor,clarithromycin,amoxicillin or metronidazole

INTERVENTIONS:
Drug: Proton pump inhibitor,clarithromycin,amoxicillin or metronidazole — Triple or quadruple therapy consist of Proton pump inhibitor,clarithromycin,amoxicillin or metronidazole.

SUMMARY:
Clarithromycin (CLA)、amoxicillin (AMO)、metronidazole (MET)、levofloxacin (LEV) and tetracycline (TET) are commonly used antibiotics for Helicobacter pylori (Hp) therapy. However, the efficacy of treatment for Helicobacter pylori infection has decreased due to increasing resistance to CLA, MET and LEV. Studies had reported that beside antibiotics resistance, other factors such as age, sex, underlying disease, etc. may also affect the treatment efficacy. In some cases, when the MIC values were beyond the breakpoint, H. pylori strains with lower MIC value had better eradication than the ones with higher MIC value. However, few study investigated the relationship between MIC values and treatment outcome.

The investigators aimed to analyze the impact of influencing factors, especially minimal inhibitory concentration (MIC) value, on the efficacy of different treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* patients (aged ≥ 20 years old) with H. pylori infection between Jan. 1994 to Mar. 2018

Exclusion Criteria:

* without antibiotics susceptible test result, without treatment outcome, history of any gastrointestinal surgery, serious concomitant (renal failure, liver cirrhosis, heart failure and disease need immunosuppressant for therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 1821 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship between eradication rate (%) of therapy regimen and influencing factors (eg. sex, age, diagnosis, MIC). | 4 weeks after treatment finished.

CONTACTS AND LOCATIONS:
Locations (1):
- Tzu-Chi Lai, Taipei, No.33, Linsen S. Rd., Zhongzheng Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No